CLINICAL TRIAL: NCT05059015
Title: Effect of HPV Self-collection in Adherence to Cervical Cancer Screening Algorithms
Brief Title: Human Papilloma Virus (HPV) Self-collection and Women Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C19010300532
Record Dates: First submitted 2021-08-12; First posted 2021-09-28 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-08

CONDITIONS: Cervical Cancer; HPV Infection
Keywords: Cervical Cancer; Screening programs; HPV tests
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial with three arms will be performed: One group with the routine screening procedure based on HPV tests with cervical sampling by a health personnel ( 3 visits: sampling, colpo/biopsy, treatment of CIN2 +), a second group with a screening based on HPV self-testing and colposcopic evaluation (2 visits: colpo/biopsy, treatment of CIN2 + ); and a third group with a screening based only on HPV self-testing (1 visit: HPV + treatment according to eligibility).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CERVICAL HPV (Active Comparator): Routine screening procedure based on HPV tests with cervical sampling by a health personnel
  Interventions: Diagnostic Test: CERVICAL HPV
- SELF SAMPLING HPV ARM 2 (Experimental): Screening based on HPV self-testing and colposcopic evaluation
  Interventions: Diagnostic Test: SELF SAMPLING HPV
- SELF SAMPLING HPV ARM 3 (Experimental): Arm 3: screening based only on HPV self-testing
  Interventions: Diagnostic Test: SELF SAMPLING HPV

INTERVENTIONS:
Diagnostic Test: CERVICAL HPV — A screening test with an HPV test is performed by a health professional plus cytology taking, if it reports positive, colposcopy and biopsy are taken, those with a CIN2 + report are directed to receive treatment.
  Arms: CERVICAL HPV
Diagnostic Test: SELF SAMPLING HPV — A screening test is performed with an HPV test by self-testing, if it reports positive, women will receive ablative treatment according to eligibility criteria. If they do not meet the criteria for ablation, they will be referred for excisional treatment.
  Arms: SELF SAMPLING HPV ARM 2; SELF SAMPLING HPV ARM 3

SUMMARY:
Despite declining mortality in high-income countries, cervical cancer continues to be a public health problem in low and middle -income countries. HPV tests have shown a better sensibility and a higher capacity of reducing mortality than cytology based-screening. Greater participation has been demonstrated with the use of HPV self-testing when it is offered to women with a poor screening history; however, it is not clear whether getting tested necessarily translates into a greater adherence to the entire clinical protocol, including diagnosis and treatment of precancerous lesions. The aim of this study is to evaluate the effect of the self-testing techniques on the participation and adherence of women to cervical cancer screening.

DETAILED DESCRIPTION:
The investigators will perform a randomized clinical trial with three arms including: regular HPV with cytology triage, colpo/biopsy, and treatment if indicated; HPV self-collection without cytology triage but with colpo/biopsy and treatment if indicated, HPV self-collection with immediate treatment for women with positive test results. This study will be carried out in two different settings with differential access to diagnosis and treatment. Two methods will be used for inviting women and collecting samples: mail and door-to-door. Participation (screening uptake) and adherence to the clinical protocol (compliance with diagnosis and treatment) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women 30-65 years old
* No history of cytology or any other screening test for cancer of the cervix in the past 5 years
* Be linked to one of the health providing entities participating in the study
* Women who sign the informed consent.

Exclusion Criteria:

* Women 30-65 years old
* No history of cytology or any other screening test for cancer of the cervix in the past 5 years
* Be linked to one of the health providing entities participating in the study
* Women who sign the informed consent.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with no history of cytology or any other screening test for cancer of the cervix in the past 5 years
Enrollment: 80 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2022-12-03 (Estimated)

PRIMARY OUTCOMES:
Participation | 1 year
  Number of women that undergo the screening test / total number of women invited.
Adherence | 1 year
  Number of women that undergo the screening test + women who completed the diagnosis and treatment process / total number of women invited + total number of women with a positive screening in follow-up protocols.

SECONDARY OUTCOMES:
Quality of HPV samples | 1 year
  Number of samples suitable for analysis / Total number of samples
CIN2 + rate in the study population | 1 year
  Number of CIN2 + diagnosed / total women screened
CIN2 + rate in population with positive screening | 1 year
  Number of CIN2 + diagnosed / total of women positive at screening

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cancerología, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Undecided